CLINICAL TRIAL: NCT02334670
Title: Evaluation of a Public Health Strategy to Improve Survival of HIV Infected Patients
Brief Title: Vietnam Cryptococcal Retention in Care Study Version 1.0
Acronym: CRICS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1U01GH000758 (NIH)
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Meningitis, Cryptococcal; Central Nervous System Fungal Infections; Central Nervous System Infections; Meningitis, Fungal
Keywords: cryptococcal meningitis; HIV; AIDS; Fluconazole
MeSH Terms: conditions — Meningitis, Cryptococcal; Central Nervous System Fungal Infections; Central Nervous System Infections; Meningitis, Fungal; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Complete blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CrAg(+) and CM(+): Patients with symptoms of CNS disease will be treated according to Vietnam national guidelines for HIV/AIDS management.
  Interventions: Drug: Fluconazole
- CrAg(+) and CM(-): Patients with CrAg(+) and without CM symptoms will be treated with high-dose fluconazole. The initial dosage of fluconazole will be 900 mg taken each day for 2 weeks. This will be followed by fluconazole 450 mg orally each day for 8 weeks. Finally, maintenance treatment with fluconazole 200mg orally each (2 tablets of 100 mg procured especially for the study) day will continue until CD4 >200 cells/µL for at least 6 months.
  Interventions: Drug: Fluconazole
- CrAg negative: Patients with CrAg negative results will be managed as other HIV positive patients according to the national guidelines
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — HIV-infected patients with CD4 ≤100 cells/μL who present for HIV care at outpatient clinics (OPCs) in Vietnam where CrAg screening is offered will be recruited into the study. Study participants will be screened for cryptococcal antigen using the Lateral Flow Assay (LFA). Those who are CrAg-positive, but have no features of central nervous system (CNS) disease, will be treated with high-dose fluconazole.

SUMMARY:
It is hypothesized that implementing plasma CrAg screening in clinics providing routine HIV care will enable identification of Vietnamese adult patients with advanced HIV (CD4 ≤100 cells/μL) who have early cryptococcal disease, enable prompt preemptive treatment with high-dose fluconazole, and improve survival.

DETAILED DESCRIPTION:
This is multicenter prospective cohort evaluation of the implementation of a cryptococcal antigen (CrAg) screening program in Vietnam. HIV-infected patients with CD4 ≤100 cells/μL who present for HIV care at outpatient clinics (OPCs) in Vietnam where CrAg screening is offered will be recruited into the study. Study participants will be screened for cryptococcal antigen using the Lateral Flow Assay (LFA) and followed up for 12 months with clinical assessments and the collection of routine and supplemental survey data. Those who are CrAg-positive, but have no features of central nervous system (CNS) disease, will be treated with high-dose fluconazole. Those with symptoms of CNS disease will be treated according to national guidelines. Survival, retention in care, and other clinical outcomes will be documented for patients who test CrAg-positive and are treated with fluconazole and those who test CrAg-negative.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Confirmed HIV infection using National Testing Algorithm
* CD4 ≤100 cells/μL
* Able to provide written informed consent

Exclusion Criteria:

* History of prior CM
* Receipt of systemic antifungal medication for more than 4 consecutive weeks within the past 6 months
* Currently taking ART or history of ART for more than 4 weeks within the past year
* Known to be currently pregnant or planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly registering and ART-naive patients with advanced HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 2612 (Estimated)
Dates: Start 2015-08-14 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Six (6) and (12) month all-cause and CM-related mortality among patients who screen CrAg-positive and CrAg-negative | Up to 12 months after recruitment
Proportion of all patients tested for plasma CrAg who have positive results | Up to 12 months after recruitment

SECONDARY OUTCOMES:
Percent of patients with HIV-related hospitalizations at 6 and 12 months | 12 months after recruitment
Percent of patients with new AIDS-defining OIs/conditions at 6 and 12 months | 12 months after recruitment
Causes of death | 12 months after recruitment
Six (6) and (12) month retention among patients who screen CrAg-positive and CrAg-negative | 12 months after recruitment
Percentage of patients with CD4≤ 100 cells/μL who are lost to follow-up or have incomplete documentation | 12 months after recruitment
% of patients with no documented clinic visit 30, 60, and 90 days after date of the scheduled clinic appointment | 12 months after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Van Kinh, MD, PhD, Principal Investigator — National Hospital for Tropical Diseases
Locations (1):
- National Hospital for Tropical Diseases, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
Please contact PI for any enquiries